CLINICAL TRIAL: NCT00748839
Title: Heparin-Induced Thrombocytopenia : Development and Validation of a Predictive Clinical Score: a Prospective Multicenter Study Under the Auspices of the French Haemostasis and Thrombosis Study Group (GEHT)in Cooperation With the French Association of Regional PharmacoVigilance Center (AFCRPV)
Brief Title: Heparin-Induced Thrombocytopenia: Development and Validation of a Predictive Clinical
Acronym: Score-TIH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Hyphen BioMed (Unknown); CIC-EC de Saint-Etienne (Unknown); Groupe d'étude sur l'Hémostase et la Thrombose (Unknown); Association Française des centres régionaux de Pharmacovigilance (Unknown); Laboratoires Organon (Unknown); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 0801016
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Heparin-induced Thrombocytopenia
Keywords: HIT; Heparin-induced thrombocytopenia; heparin treatment; venous thrombosis; arterial thrombosis; predictive clinical score; biological test; anti-H-PF4 antibodies
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Although Heparin-induced thrombocytopenia (HIT) is a rare complication of heparin treatment, it results in a high rate of morbidity and mortality, the cumulative rate of thrombosis recurrence, amputation and death approaching 52 % at one month if no specific treatment is initiated. It is therefore vital to diagnose HIT as early and as reliably as possible to permit appropriate management of this rare condition.

During the acute phase of HIT, clinicians and biologists can only suspect this complication with a greater or lesser degree of confidence. Clinical data are not sufficiently sensitive or specific to confirm or refute thr diagnosis of HIT.

DETAILED DESCRIPTION:
Purpose : To create and validate a score predicting the diagnosis of HIT

ELIGIBILITY:
Inclusion Criteria:

* all patients presenting, either during or immediately after treatment:

  * thrombocytopenia and/or venous or arterial thrombosis
  * for whom a request for biological assessment to check for HIT (anti-H-PF4 ELISA test) is to be addressed to the specialized haemostasis laboratory participating in the study

Exclusion Criteria:

* do not possess sufficient clinical data prior to performance of the biological test
* cannot assure follow-up of the patient until normalization of the platelet count

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
the final diagnosis of HIT established by five independent experts in haemostasis and determined by thrombocytopenia and confirmation of HIT by immunological and/or functional tests | inclusion and 40 days after the inclusion

SECONDARY OUTCOMES:
pathogenic nature of anti HPF4 antibodies of IgM and IgA type | inclusion
new biological test detecting HIT | inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Bernard TARDY, MD, Principal Investigator — CHU de Saint-Etienne
Locations (27):
- France (27):
  - ETS de Franche Conté - Laboratoire d'Immuno Hématologie, Besançon
  - CHU Cavale Blanche Laboratoire d'Hématologie, Brest
  - Laboratoire d'hématologie - Hôpital Louis Pradel, Bron
  - Hôpital Antoine Beclère - Laboratoire d'hématologie, Clamart
  - Laboratoire d'hématologie - CHU de Clermont Ferrand, Clermont-Ferrand
  - HCC Colmar - laboratoire d'hématologie, Colmar
  - Laboratoire d'Hématologie - CHU le Bocage, Dijon
  - Laboratoire d'hémostase - CCML, Le Plessis-Robinson
  - Hôpital Cardiologique - Laboratoire d'Hémostase, Lille
  - CHU La Timone - Laboratoire Hématologie, Marseille
  - Hôpital SAINT ELOI - CHU de Montpellier - Laboratoire d'Hématologie, Montpellier
  - Hématologie biologique - CHU Nancy, Nancy
  - HOTEL DIEU - CHU Nantes - Laboratoire d'Hématologie, Nantes
  - Hématologie Biologique - Hôpital Tenon,, Paris
  - Hôpital Necker Enfants Malades -Laboratoire d'Hématologie, Paris
  - Hôpital BICHAT - Service d'hématologie immunologie, Paris
  - G.H. Pitié Salpétrière - Labo Hémostase Pavillon Laveran, Paris
  - Hôpital Européen Georges Pompidou - Service Hématologie Biologique A, Paris
  - Hôpital Cardiologique - CHU Bordeaux, Pessac
  - Laboratoire central d'hématologie - Hôpital R. DEBRE, Reims
  - CHU de ROUEN, Rouen
  - Laboratoire d'hématologie, Saint-Etienne
  - Service d'Urgence et de Réanimation, Saint-Etienne
  - CHU Strasbourg Hautepierre Laboratoire d'Hématologie, Strasbourg
  - CMC Foch Laboratoire d'hémostase, Suresnes
  - Hopital Purpan - Laboratoire d'hématologie, Toulouse
  - CHU Trousseau - CTH - Service d'Hématologie Hémostase, Tours

REFERENCES:
- [Derived] Tardy-Poncet B, de Maistre E, Pouplard C, Presles E, Alhenc-Gelas M, Lasne D, Horellou MH, Mouton C, Serre-Sapin A, Bauters A, Nguyen P, Mullier F, Perrin J, Le Gal G, Morange PE, Grunebaum L, Lillo-Le Louet A, Elalamy I, Gruel Y, Greinacher A, Lecompte T, Tardy B; GFHT-HIT study group. Heparin-induced thrombocytopenia: Construction of a pretest diagnostic score derived from the analysis of a prospective multinational database, with internal validation. J Thromb Haemost. 2021 Aug;19(8):1959-1972. doi: 10.1111/jth.15344. Epub 2021 Jun 14. PMID 33872452